CLINICAL TRIAL: NCT02980523
Title: A Randomized, Double Blind, Phase II Multicenter Trial to Evaluate the Safety and Efficacy of PRO-157 Ophthalmic Solution in Three Different Dosing Regimen Versus Moxifloxacin Versus Gatifloxacin in Patients With Bacterial Conjunctivitis.
Brief Title: Safety and Efficacy of PRO-157 vs Moxifloxacin vs Gatifloxacin in Patients With Bacterial Conjunctivitis (Pazufloxacin)
Acronym: Pazufloxacin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH157-0114/II
Record Dates: First submitted 2016-11-17; First posted 2016-12-02 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — pazufloxacin; Ophthalmic Solutions; Moxifloxacin; Gatifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PRO-157 BID (2 times per day) (Experimental): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 12 hours per day (BID), for 7 days
  2. instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%)every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  Interventions: Drug: PRO-157; Drug: Lagricel Ofteno®
- PRO-157 TID (3 times per day) (Experimental): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 8 hours per day (TID), for 7 days
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  Interventions: Drug: PRO-157; Drug: Lagricel Ofteno®
- PRO-157 QID (4 times per day) (Experimental): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 6 hours per day (QID), for 7 days
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  Interventions: Drug: PRO-157; Drug: Lagricel Ofteno®
- Moxifloxacin (Vigamox®) (Active Comparator): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of Moxifloxacin, every 8 hours per day, for 7 days.
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day for 7 days. (Can be applied 15 minutes after moxifloxacin)
  Interventions: Drug: Vigamox; Drug: Lagricel Ofteno®
- Gatifloxacin (Zymar®) (Active Comparator): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of Gatifloxacin, every 8 hours per day, for 7 days.
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day for 7 days.one drop 4 times a day for 7 days in each eye.(Can be applied 15 minutes after gatifloxacin)
  Interventions: Drug: Zymar®; Drug: Lagricel Ofteno®

INTERVENTIONS:
Drug: PRO-157 — PRO-157 (Pazufloxacin 0.06%) Laboratories Sophia S.A. de C.V., ophthalmic solution
  Other Names: Pazufloxacin 0.06%, ophthalmic solution
  Arms: PRO-157 BID (2 times per day); PRO-157 QID (4 times per day); PRO-157 TID (3 times per day)
Drug: Vigamox — Vigamox® (Moxifloxacin 0.5%), Alcon Laboratories, S.A. de C.V., ophthalmic solution
  Other Names: Moxifloxacin
  Arms: Moxifloxacin (Vigamox®)
Drug: Zymar® — Zymar® (Gatifloxacin 0.3%), Allergan, S.A. de C.V., ophthalmic solution
  Other Names: Gatifloxacin
  Arms: Gatifloxacin (Zymar®)
Drug: Lagricel Ofteno® — Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
  Other Names: Sodium hyaluronate 0.4%

SUMMARY:
A randomized, double blind, phase II multicenter trial with the objective of assess the safety and efficacy of the PRO-157 ophthalmic solution in three different dosing regimens, versus Moxifloxacin, versus Gatifloxacin in patients with bacterial conjunctivitis.

Number of participants: 300 eyes, 60 per group.

Criteria for evaluation:

Measurements of effectiveness: Main efficacy criterion It will be determined as effective if there is a reduction in number or species of bacterial flora by comparing the basal culture against the final culture among the five different patient groups.

Reduction or absence of infection with the clinical evaluation through signs and symptoms.

Safety Measurements: it will be determined by visual acuity and adverse events Patients recruited will be treated for 7, for protocol purpose, the infected eye (s) will be taken into account at the time of baseline, however the study medication and procedures will be applied and performed in both eyes to protect the healthy eye.

The study is divided into the following evaluation periods:

Visit 1 baseline (day 1), visit 2 (day 3), final visit (day 8) and a telephone call (day 23) for the evaluation of adverse events.

Subjects will be allocated to any of the following regimen dosages:

* PRO-157 1 drop 2 times daily
* PRO-157 1 drop 3 times daily
* PRO-157 1 drop 4 times daily
* Moxifloxacin 1 drop 3 times daily
* Gatifloxacin 1 drop 3 times daily. All regimen dosage will have a duration of 7 days. An artificial tear preservative free (Lagricel Ofteno®) will also be applied 15 minutes before instillation of study drug, during study period.

Data Analysis: The data will be analyzed by Intention to Treat (ITT) and per Protocol (PP) in which each of the variables is described, the ITT population will be constituted by all subjects recruited who have received at least one dose of the study, the PP population will be the subset of ITT composed of all subjects without any major deviation from the protocol and the bivariate analysis will be performed in this group.

Continuous quantitative variables are expressed and presented by measures of central tendency and dispersion (mean, standard deviation and ranges). Qualitative nominal and ordinal variables are presented by means of frequencies and proportions. The level of significance was an alpha of 0.05 or less.

DETAILED DESCRIPTION:
Lagricel Ofteno® is a registered trademark, therefore the use of the same throughout the document can not be translated into the English language.

PRO-157, the acronym is part of an internal code used to record formulations or research projects and the numbers indicate consecutive of the molecule under study.

ELIGIBILITY:
Inclusion Criteria:

* Obtained from physician office visit.
* Diagnosis of bacterial conjunctivitis (signs and / or symptoms and / or culture).
* Informed Consent signed and dated (consent of the parents for minor patients).

Exclusion Criteria:

* absence of written informed consent.
* Women of childbearing age, without contraceptive use (oral contraceptive pill, contraceptive intrauterine device, contraceptive implant, patch or condom).
* Pregnant or breastfeeding women.
* Subjects that could not be evaluated partially or totally according to the protocol.
* Subjects with topical, systemic or intravenous medication with any type of antibiotic on the day of the baseline visit.
* Subjects with topical, systemic or intravenous medication with any type of medication that interferes decisively with the results of the study.
* Subjects with a hypersensitivity history to any component or analogues of the formulation product.
* Positive drug addiction (smoking, alcoholism, marijuana).
* Subjects with a history of participation in any clinical study in the last 40 days prior to their evaluation.
* incapacity to give informed consent owing to mental disorder or legal condition.
* Any major anomaly detected during the clinical examination, tests that could interfere with the performance of the study or with the efficacy and safety evaluations.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza, MD, Study Director — Laboratorios Sophia
Locations (1):
- Unidad Medica "Grupo Pediátrico", Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- PRO-157 BID (2 Times Per Day): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 12 hours per day (BID), for 7 days
  2. instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%)every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  PRO-157: PRO-157 (Pazufloxacin 0.09%) Laboratories Sophia S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
- PRO-157 TID (3 Times Per Day): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 8 hours per day (TID), for 7 days
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  PRO-157: PRO-157 (Pazufloxacin 0.09%) Laboratories Sophia S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
- PRO-157 QID (4 Times Per Day): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 6 hours per day (QID), for 7 days
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  PRO-157: PRO-157 (Pazufloxacin 0.09%) Laboratories Sophia S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
- Moxifloxacin (Vigamox®): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of Moxifloxacin, every 8 hours per day, for 7 days.
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day for 7 days. (Can be applied 15 minutes after moxifloxacin)
  Vigamox: Vigamox® (Moxifloxacin 0.5%), Alcon Laboratories, S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
- Gatifloxacin (Zymar®): 60 eyes of 30 research subjects will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of Gatifloxacin, every 8 hours per day, for 7 days.
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day for 7 days.one drop 4 times a day for 7 days in each eye.(Can be applied 15 minutes after gatifloxacin)
  Zymar®: Zymar® (Gatifloxacin 0.3%), Allergan, S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
Period: Overall Study
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Started | 30; 60 eyes | 30; 60 eyes | 30; 60 eyes | 30; 60 eyes | 30; 60 eyes
Completed | 27; 54 eyes | 19; 38 eyes | 24; 48 eyes | 21; 42 eyes | 20; 40 eyes
Not Completed | 3; 6 eyes | 11; 22 eyes | 6; 12 eyes | 9; 18 eyes | 10; 20 eyes
Not completed — Lost to Follow-up | 1 | 4 | 1 | 2 | 1
Not completed — Excluded from analysis | 1 | 3 | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 4 | 4 | 5 | 8
Not completed — Did not receive intervention | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- PRO-157 BID: One drop twice a day for 7 days (PRO-157=pazufloxacin 0.6%)
- PRO-157 TID; PRO-157 QID: One drop three times a day for 7 days (PRO-157=pazufloxacin 0.6%)
- Moxifloxacine: One drop four times a day for 7 days Moxifloxacin 0.5% (Vigamox®).
- Gatifloxacine: One drop four times a day for 7 days Gatifloxacin 0.3% (Zymar®).
- Total: Total of all reporting groups
Arm/Group | PRO-157 BID | PRO-157 TID | PRO-157 QID | Moxifloxacine | Gatifloxacine | Total
Number analyzed (Participants) | 27 | 19 | 24 | 21 | 20 | 111
Number analyzed (eyes) | 54 | 38 | 48 | 42 | 40 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 7 | 5 | 5 | 27
  Between 18 and 65 years | 11 | 13 | 10 | 11 | 8 | 53
  >=65 years | 9 | 3 | 7 | 5 | 7 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (27.9) | 37.2 (21.3) | 43.3 (25.7) | 39.9 (26.9) | 43.4 (29.5) | 40.8 (26.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 16 | 13 | 11 | 69
  Male | 8 | 9 | 8 | 8 | 9 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico: Mexicans | 27 | 19 | 24 | 21 | 20 | 111
  Mexico: others | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Bacterial Culture
Description: Efficacy will be determined comparing the cultures of the lower conjunctival pouch, of the baseline (day 1) against final visit (day 8), quantifying and identifying the colony forming units (CFU) by genus and species.
  The evaluated variable is discrete quantitative type and the scale of measurement used will be CFU x mL considering the eradication, reduction or proliferation of the bacterial agent. It will be determined as effective if there is a reduction in number of bacterial flora in at least 95% of the evaluated subjects.
Time Frame: up to one week
Population: Treatment analysis, a culture was performed per eye
Measure: Number; unit: cultures
Units Other Than Participants: cultures
Groups:
- Moxifloxacin (Vigamox®): 60 eyes will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of Moxifloxacin, every 8 hours per day, for 7 days.
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day for 7 days. (Can be applied 15 minutes after moxifloxacin)
  Vigamox: Vigamox® (Moxifloxacin 0.5%), Alcon Laboratories, S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
- Gatifloxacin (Zymar®): 60 eyes will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of Gatifloxacin, every 8 hours per day, for 7 days.
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day for 7 days.one drop 4 times a day for 7 days in each eye.(Can be applied 15 minutes after gatifloxacin)
  Zymar®: Zymar® (Gatifloxacin 0.3%), Allergan, S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Number analyzed (Participants) | 15 | 8 | 13 | 15 | 9
Number analyzed (cultures) | 30 | 16 | 26 | 29 | 17
cultures
  basal cultures positives | 30 | 16 | 26 | 29 | 17
  final cultures negatives | 17 | 14 | 16 | 28 | 15
Statistical Analysis 1: Comparison: PRO-157 BID (2 Times Per Day) vs PRO-157 TID (3 Times Per Day) vs PRO-157 QID (4 Times Per Day) vs Moxifloxacin (Vigamox®) vs Gatifloxacin (Zymar®); Test type: Non-Inferiority or Equivalence — The aim of this study was to find the ideal dose of treatment for bacterial eradication and non-inferiority with the comparative groups; p = 0.002, Chi-squared

2. Primary Outcome: Adverse Events
Description: Number of adverse events: dependent variable, discrete quantitative, the number of adverse events per group will be compared at the end of the study and it will be considered safe if there is not greater increase of 5% of serious adverse events.
Time Frame: during the intervention period for 7 days, and 15 days after the final visit
Population: Treatment analysis
Measure: Number; unit: events
Units Other Than Participants: eyes
Groups:
- PRO-157 BID (2 Times Per Day): 60 eyes will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 12 hours per day (BID), for 7 days
  2. instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%)every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  PRO-157: PRO-157 (Pazufloxacin 0.09%) Laboratories Sophia S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
- PRO-157 TID (3 Times Per Day): 60 eyes will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 8 hours per day (TID), for 7 days
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  PRO-157: PRO-157 (Pazufloxacin 0.09%) Laboratories Sophia S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
- PRO-157 QID (4 Times Per Day): 60 eyes will be evaluated with the following therapeutic regimen:
  1. instill one drop in each eye of PRO-157 (pazufloxacin), every 6 hours per day (QID), for 7 days
  2. 15 minutes after, instill one drop in each eye of Lagricel Ofteno® (Sodium hyaluronate 0.4%) every 6 hours per day, for 7 days. (Can be applied 15 minutes after PRO 157)
  PRO-157: PRO-157 (Pazufloxacin 0.09%) Laboratories Sophia S.A. de C.V., ophthalmic solution
  Lagricel Ofteno®: Lagricel Ofteno® Sodium hyaluronate 0.4%, Laboratories Sophia S.A. de C.V., ophthalmic solution
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Number analyzed (Participants) | 27 | 19 | 24 | 21 | 20
Number analyzed (eyes) | 54 | 38 | 48 | 42 | 40
events | 7 | 5 | 7 | 4 | 7
Statistical Analysis 1: Comparison: PRO-157 BID (2 Times Per Day) vs PRO-157 TID (3 Times Per Day) vs PRO-157 QID (4 Times Per Day) vs Moxifloxacin (Vigamox®) vs Gatifloxacin (Zymar®); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.372, Chi-squared, Corrected

3. Secondary Outcome: Cases Frequency of Ocular Secretion
Description: Secretion ocular: qualitative ordinal variable. The secretion was evaluated by subject of study as present / absent, taking into consideration that each study subject represents two probable cases, one for each eye. On this premise, the statistical analysis of the number of cases reported in the final visit was made by study group.
Time Frame: Up to one week.
Population: treatment analysis.
Measure: Number; unit: secretion cases reported
Units Other Than Participants: eyes
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Number analyzed (Participants) | 27 | 19 | 24 | 21 | 20
Number analyzed (eyes) | 54 | 38 | 48 | 42 | 40
secretion cases reported | 0 | 3 | 0 | 7 | 2
Statistical Analysis 1: Comparison: PRO-157 BID (2 Times Per Day) vs PRO-157 TID (3 Times Per Day) vs PRO-157 QID (4 Times Per Day) vs Moxifloxacin (Vigamox®) vs Gatifloxacin (Zymar®); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.341, Chi-squared, Corrected

4. Secondary Outcome: Number of Cases of Conjunctival Hyperemia
Description: Conjunctival hyperemia: qualitative ordinal variable. The conjunctival hyperemia was evaluated by subject of study as present / absent, taking into consideration that each study subject represents two probable cases, one for each eye. On this premise, the statistical analysis of the number of cases reported in the final visit was made by study group.
Time Frame: up to one week
Population: Treatment analysis
Measure: Number; unit: hyperemia cases reported
Units Other Than Participants: eyes
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Number analyzed (Participants) | 27 | 19 | 24 | 21 | 20
Number analyzed (eyes) | 54 | 38 | 48 | 42 | 40
hyperemia cases reported | 17 | 1 | 5 | 7 | 8
Statistical Analysis 1: Comparison: PRO-157 BID (2 Times Per Day) vs PRO-157 TID (3 Times Per Day) vs PRO-157 QID (4 Times Per Day) vs Moxifloxacin (Vigamox®) vs Gatifloxacin (Zymar®); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.001, Chi-squared, Corrected

5. Secondary Outcome: Chemosis Frequency
Description: Chemosis: qualitative ordinal variable, measurement scale absent or present. The chemosis was evaluated by subject of study as present / absent, taking into consideration that each study subject represents two probable cases, one for each eye. On this premise, the statistical analysis of the number of cases reported in the final visit was made by study group.
Time Frame: up to one week
Population: Treatment analysis
Measure: Number; unit: chemosis cases reported
Units Other Than Participants: eyes
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Number analyzed (Participants) | 27 | 19 | 24 | 21 | 20
Number analyzed (eyes) | 54 | 38 | 48 | 42 | 40
chemosis cases reported | 0 | 0 | 0 | 6 | 2
Statistical Analysis 1: Comparison: PRO-157 BID (2 Times Per Day) vs PRO-157 TID (3 Times Per Day) vs PRO-157 QID (4 Times Per Day) vs Moxifloxacin (Vigamox®) vs Gatifloxacin (Zymar®); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.003, Chi-squared, Corrected

6. Secondary Outcome: Eyelid Edema Frequency
Description: Eyelid edema: qualitative ordinal variable, measurement scale absent or present.Between baseline (day 0) versus final visit (day 7).
  The eyelid edema was evaluated by subject of study as present / absent, taking into consideration that each study subject represents two probable cases, one for each eye. On this premise, the statistical analysis of the number of cases reported in the final visit was made by study group.
Time Frame: Up to one week
Population: Treatment analysis
Measure: Number; unit: eyelid edema cases reported
Units Other Than Participants: eyes
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Number analyzed (Participants) | 27 | 19 | 24 | 21 | 20
Number analyzed (eyes) | 54 | 38 | 48 | 42 | 40
eyelid edema cases reported | 6 | 0 | 4 | 4 | 6
Statistical Analysis 1: Comparison: PRO-157 BID (2 Times Per Day) vs PRO-157 TID (3 Times Per Day) vs PRO-157 QID (4 Times Per Day) vs Moxifloxacin (Vigamox®) vs Gatifloxacin (Zymar®); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.216, Chi-squared, Corrected

7. Secondary Outcome: Frequency of Corneal Epithelial Defects
Description: Corneal epithelial defects: qualitative ordinal variable, measurement scale present or absent.
  The corneal epithelial defects was evaluated by subject of study as present / absent, taking into consideration that each study subject represents two probable cases, one for each eye. On this premise, the statistical analysis of the number of cases reported in the final visit was made by study group.
Time Frame: Up to one week
Population: Treatment analysis
Measure: Number; unit: Corneal defects cases reported
Units Other Than Participants: eyes
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Number analyzed (Participants) | 27 | 19 | 24 | 21 | 20
Number analyzed (eyes) | 54 | 38 | 48 | 42 | 40
Corneal defects cases reported | 9 | 4 | 6 | 5 | 5
Statistical Analysis 1: Comparison: PRO-157 BID (2 Times Per Day) vs PRO-157 TID (3 Times Per Day) vs PRO-157 QID (4 Times Per Day) vs Moxifloxacin (Vigamox®) vs Gatifloxacin (Zymar®); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.829, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the intervention period for 8 days, and a follow-up call was made 15 days after the final visit.
Description: Adverse events were recorded according to the patient's scheduled or unscheduled visits, and were given a diary in which they could make annotations of their symptoms, the investigator reviewed these symptoms and reported on them The format of adverse events.
Arm/Group | PRO-157 BID (2 Times Per Day) | PRO-157 TID (3 Times Per Day) | PRO-157 QID (4 Times Per Day) | Moxifloxacin (Vigamox®) | Gatifloxacin (Zymar®)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 7/30 | 5/30 | 7/30 | 3/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-157 BID (2 Times Per Day) (N=30) | PRO-157 TID (3 Times Per Day) (N=30) | PRO-157 QID (4 Times Per Day) (N=30) | Moxifloxacin (Vigamox®) (N=30) | Gatifloxacin (Zymar®) (N=30)
urinary tract infection (ITU) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ischemic optic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-157 BID (2 Times Per Day) (N=30) | PRO-157 TID (3 Times Per Day) (N=30) | PRO-157 QID (4 Times Per Day) (N=30) | Moxifloxacin (Vigamox®) (N=30) | Gatifloxacin (Zymar®) (N=30)
Eyelid ecchymosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
stomach flu (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hordeolum (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Numular keratitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lack of effectiveness (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritant conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Systemic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Preseptal cellulitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
stomachache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In the present study the efficacy of pazufloxacin at different doses has not been demonstrated. In addition, the minimum inhibitory dose for ophthalmic administration is not established. Cultures could also not be determined in all study subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI (s) can not make use of the partial or total information of this investigation, due to the clauses contained in the agreement of confidentiality of the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT02980523/Prot_SAP_000.pdf